CLINICAL TRIAL: NCT01291030
Title: The Impact of Magnesium Supplementation on Insulin Resistance and Secretion in Renal Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010/416
Record Dates: First submitted 2011-02-04; First posted 2011-02-07 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Glucose Metabolism; Renal Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- hypomagnesemic + magnesium supplement (Experimental): The patient group of hypomagnesesemic renal transplant recipients randomized to magnesium supplementation (number = 30). The assessments are a baseline fasting assessment of insulin resistance and an Oral Glucose Tolerance Test with derived indices of insulin secretion,which are repeated after 6 months.
  Interventions: Dietary Supplement: magnesium supplementation
- hypomagnesemic without magnesium supplement (No Intervention): The patient group of hypomagnesesemic renal transplantation recipients, randomized to no magnesium supplementation (number = 30). During 6 months, no magnesium supplementation is started, provided that the serum magnesium level remains > 1,2 milligram/deciliter. In case of cramps, intermittent supplementation is allowed, but will be recorded. The assessments are a baseline fasting assessment of insulin resistance and an Oral Glucose Tolerance Test with derived indices of insulin secretion,which are repeated after 6 months.
- normomagnesemic without magnesium supplement (No Intervention): In the control group of normomagnesemic renal transplantation recipients (number = 10), only a baseline assessment will be performed. The assessments are a baseline fasting assessment of insulin resistance and an Oral Glucose Tolerance Test with derived indices of insulin secretion.

INTERVENTIONS:
Dietary Supplement: magnesium supplementation — The supplementation starts with 450 mg of magnesium oxide daily, up to a maximum of 3 times 450 mg daily, while aiming at a serum magnesium level of > 1,9 mg/dl.
  Arms: hypomagnesemic + magnesium supplement

SUMMARY:
Hypomagnesemia is common in renal transplant recipients and is mainly because of enhanced renal magnesium wasting, caused by immunosuppressive drugs (calcineurin inhibitors). Glucose metabolism disorders, including insulin resistance and decreased insulin secretion, are also prevalent post-transplantation and often precede the development of diabetes. As magnesium supplementation has been demonstrated to increase insulin sensitivity in both diabetic and non-diabetic patients, its potential therapeutic supplementation (post-transplantation) deserves further examination. The hypothesis is that magnesium supplementation in renal transplant recipients exerts a beneficial effect on insulin resistance and/or secretion.

ELIGIBILITY:
Inclusion Criteria:

* Renal transplantation recipients
* > 18 years of age
* more than 4 months post-transplantation
* Hypomagnesemia < 1,8 milligram/deciliter on 2 consecutive blood samples (laboratory reference interval 1,7 - 2,55 milligram/deciliter) at least 1 month apart.

Exclusion Criteria:

* Pre-existing diabetes mellitus defined as the intake of anti-diabetic drugs at the time of inclusion
* Biopsy that proves acute rejection and consecutive treatment with corticosteroid boluses less than 2 months before inclusion
* Serum creatinine > 3 milligram/deciliter
* Active infection (C reactive protein > 3 milligram/deciliter)
* Severe hypomagnesemia (< 1,2 milligram/deciliter)
* Hypokalemia (< 3,5 milli-equivalent/liter)
* Severe hypocalcemia (< 6,5 milligram/deciliter)
* Intake of digoxin
* Intake of magnesium supplementation up to 2 weeks before randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of change in insulin resistance/secretion | after 6 months
  The primary outcome of the study is the evaluation of change in insulin resistance and insulin secretion after 6 months of supplementation (versus no supplementation). Insulin resistance is measured by 'Homeostatic Model Assessment' (HOMA) - modeling and the McAuley Index. Insulin secretion is assessed by 'Oral Glucose Tolerance test' (OGTT)- derived indices.

SECONDARY OUTCOMES:
Evaluation of change in Hemoglobin A1c (HbA1C) | after 6 months
  The secondary outcome is the evaluation of change in Hemoglobin A1c after 6 months of magnesium supplementation versus no supplementation.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Van Laecke, MD, Principal Investigator — University Hospital, Ghent
Locations (2):
- Belgium (2):
  - OLV Aalst, Aalst
  - University Hospital Ghent, Ghent

REFERENCES:
- See also: Related Info — http://www.uzgent.be